CLINICAL TRIAL: NCT02925832
Title: Comparison Between Ropivacaine and Bupivacaine in Deep Topical Fornix Nerve Block Anesthesia in Patients Undergoing Cataract Surgery by Phacoemulsification.
Brief Title: Comparing Ropivacaine and Bupivacaine in DTFNB Anesthesia in Patients Undergoing Phacoemulsification
Acronym: DTFNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Dr Rahul Varshney, Post Graduate, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 273/IEC/R-26.08.2016
Record Dates: First submitted 2016-09-30; First posted 2016-10-06 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cataract Unilateral Pending Extraction; Anesthesia
Keywords: Deep topical fornix nerve block Anesthesia; Ropivacaine; Bupivacaine; Anaesthesia; Eye surgery blocks; Phacoemulsification
MeSH Terms: interventions — Ropivacaine; Anesthesia, Local; Bupivacaine; proxymetacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Experimental): Deep Topical Fornix Nerve block anesthesia using bupivacaine and proparacaine
  Interventions: Procedure: Deep Topical Fornix Nerve block anesthesia; Drug: Bupivacaine; Drug: Proparacaine
- Group R (Experimental): Deep Topical Fornix Nerve block anesthesia using ropivacaine and proparacaine
  Interventions: Procedure: Deep Topical Fornix Nerve block anesthesia; Drug: Ropivacaine; Drug: Proparacaine

INTERVENTIONS:
Procedure: Deep Topical Fornix Nerve block anesthesia — DTFNB would be performed using two sponges (2x3mm) soaked with either 0.5% bupivacaine or 0.75% ropivacaine, applied deep in the conjunctival fornices after anaesthetising the conjunctiva with proparacaine local anaesthetic drops. The sponges are to be removed after 15 minutes.
  Other Names: DTFNB
Drug: Ropivacaine — 0.75% ropivacaine soaked sponges
  Other Names: Local anaesthetic
  Arms: Group R
Drug: Bupivacaine — 0.5% bupivacaine soaked sponges
  Other Names: Local anaesthetic
  Arms: Group B
Drug: Proparacaine — For anaesthetising conjunctiva
  Other Names: Local anesthetic

SUMMARY:
Deep topical fornix nerve block anaesthesia is now a known form of nerve block for cataract surgeries by phacoemulsification. In this study the investigators intend to compare ropivacaine and bupivacaine in various parameters during phacoemulsification.

DETAILED DESCRIPTION:
Prospective, study will be conducted on 100 patients undergoing elective cataract surgery by phacoemulsification under Deep topical fornix nerve block at Government medical college, Haldwani, India.

Written informed consent to participate in the study will be taken from all the patients.

Patients will be randomly allocated into two groups, Groups B (Bupivacaine: n=50) and Group R (Ropivacaine: n =50).

Deep topical fornix nerve block (DTFNB) would be performed using two sponges (2x3 mm) soaked with either 0.5% bupivacaine or 0.75% ropivacaine, applied deep in the conjunctival fornices after anesthetizing the conjunctiva with proparacaine local anesthetic drops. The sponges are to be removed after 15-20 minutes. The anesthetic effect will be tested by grasping the limbus with Castroviejo 0.12 tissue forceps. No sedative systemic medications will be given to patients perioperatively.

All surgeries will be performed by the same surgeon. Both patients and surgeon will be blind to which anesthetic agent would be used. A 2.8mm scleral tunnel incision will be made, followed by capsulorhexis. The nucleus would be removed by the stop and chop technique followed by irrigation aspiration of the cortex. Foldable acrylic intraocular lens would be implanted in the capsular bag followed by wash of the viscoelastic and hydration of the side ports.

A simple pain scoring system will be used during the surgery (0: No pain; 1: Discomfort; 2: Pain). Assessment will be made by verbally asking the patient to score each step of the surgery i.e. scleral tunnel Incision, capsulorhexis, hydrodissection, phacoemulsification, irrigation aspiration, intraocular lens implantation and stromal hydration.

In case the score being 0 or 1 no intervention will be done. But in cases of score being 2 at any stage of the surgery, an intracameral injection of 1% preservative free lignocaine will be given.

ELIGIBILITY:
Inclusion Criteria:

- Anaesthesiologists Physical Status classification system (ASA I-II) to undergo planned cataract surgery by phacoemulsification.

Exclusion Criteria:

* Younger than 50 years,
* Had any psychiatric illness (including significant anxiety),
* Nystagmus,
* Insufficient pupil dilatation,
* Very hard cataracts (NS 4-5),
* Allergy to local anaesthetics,
* Inability to understand language or
* Patient refuses the topical anaesthesia technique

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measure level of pain and discomfort during surgery | 1 hours
  A simple pain scoring system will be used during the surgery (0: No pain; 1: Discomfort; 2: Pain).
  Assessment will be made by verbally asking the patient to score each step of the surgery i.e. scleral tunnel incision, capsulorhexis, hydrodissection, phacoemulsification, irrigation aspiration, intraocular lens implantation and stromal hydration

SECONDARY OUTCOMES:
Number of patients where Supplemental anaesthesia was given | 1 hour
  Pain score being 2 at any stage of the surgery, an intracameral injection of 1% preservative free lignocaine will be given.
Level of surgeon satisfaction | 1 hour
  0: Poor,
  1. Adequate,
  2. Good
Incidence of Surgical complications | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Govind S Titiyal, Professor, Study Chair — Head of department Ophthalmology
Locations (1):
- Government medical college, Haldwani, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided